CLINICAL TRIAL: NCT06025383
Title: 2 Weeks of L-Citrulline Supplementation Improves Arterial Function and Systolic Blood Pressure at Rest and During Exercise in Postmenopausal Women With Elevated Blood Pressure and Hypertension
Brief Title: 2 Weeks of Citrulline Supplementation on Arterial Function in Postmenopausal Women With Elevated Blood Pressure or Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Arturo Figueroa, Principal Investigator, Texas Tech University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB2022-1055
Record Dates: First submitted 2023-08-19; First posted 2023-09-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2023-08

CONDITIONS: Menopause; Hypertension
Keywords: Endothelial function; Blood flow; Blood pressure; Functional sympatholysis
MeSH Terms: conditions — Hypertension | interventions — Citrulline

STUDY DESIGN:
Intervention Model Description: Cross-Over Assignment Double (Participant, Investigator) randomized, double-blind, placebo-controlled, cross-over study design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-Citrulline (Experimental): L-Citrulline: 6 grams/day divided in 2 equal doses
  Interventions: Dietary Supplement: L-Citrulline
- Placebo (Placebo Comparator): Microcrystalline cellulose: 8 capsules/day divided into 2 equal doses
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-Citrulline — 2 weeks of L-Citrulline supplementation (6 grams/day)
  Arms: L-Citrulline
Dietary Supplement: Placebo — 2 weeks of microcrystalline cellulose supplementation (8 capsules/day)
  Arms: Placebo

SUMMARY:
The objective of this project is to elucidate the effect of L-Citrulline (L-CIT) supplementation on vascular function at rest and during rhythmic handgrip exercise and functional sympatholysis via lower-body negative pressure in postmenopausal women with elevated blood pressure and hypertension.

DETAILED DESCRIPTION:
Using a double-blind, randomized, placebo-controlled, and crossover design, overweight or obese postmenopausal women with elevated blood pressure (BP) or hypertension will receive CIT (6 grams/day) or placebo for 2 weeks, separated by a two-week washout period.

There will be a total of 5 laboratory visits. The 1st visit will take approximately 1 hour. The 2nd - 5th visits will take about 2 hours and 15 minutes. Visit 1 will be a screening visit, visits 2 and 4 will be considered baseline visits, and visits 3 and 5 will be following the participants' two weeks of supplementation. Arterial stiffness (carotid-femoral and femoral-dorsalis pedis pulse wave velocity) and endothelial function will be assessed at rest. Additionally, brachial artery blood flow, forearm muscle oxygenation, cardiovascular hemodynamics (stroke volume, cardiac output, systemic vascular resistance), and BP will be assessed at rest, during 6 minutes of rhythmic handgrip exercise at 30% of a predetermined maximal voluntary contraction, and 2 minutes of superimposed lower body negative pressure to increase sympathetic activity.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (defined as the absence of menstruation for at least 1 year).
* Resting systolic blood pressure 120-150 mmHg.
* Between the ages of 50 - 70 years.
* Sedentary (< 120 minutes of exercise/week).
* Body mass index of 25 - 39.9 kg/m2.
* Fasting glucose < 126 mg/dL and HbA1c < 6.5%.

Exclusion Criteria:

* Body mass index ≥ 40 or < 25 kg/m2.
* Systolic blood pressure > 150 mmHg.
* Taking more than two antihypertensive medications.
* Cardiovascular diseases, type I/II diabetes, musculoskeletal disorders, or cancer.
* Changes in hypertensive medication in the past three months.
* Began or changed hormone replacement therapy in the past 6 months.
* Current smoker.
* Heavy drinking (> 7 alcoholic drinks/week).
* Participants on beta-blockers or other vasodilatory supplements (nitrates).
* Incorporated in a weight loss program and/or aerobic or resistance training program.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Macrovascular endothelial function at rest | 2 weeks of each intervention
  Endothelial function will be assessed via brachial artery flow-mediated vasodilation (ultrasonography) during reactive hyperemia at baseline and after 2 weeks of each supplementation.
Microvascular endothelial function at rest | 2 weeks of each intervention
  Endothelial function will be assessed via peripheral arterial tonometry (endoPAT) during reactive hyperemia at baseline and after 2 weeks of each supplementation.
Microvascular endothelial function at rest | 2 weeks of each intervention
  Endothelial function will be assessed using forearm muscle oxygen saturation (near-infrared spectroscopy) during reactive hyperemia before and after 2 weeks of each supplementation.
Brachial artery blood flow at rest and during rhythmic handgrip exercise with and without lower-body negative pressure | 2 weeks of each intervention
  Blood flow will be measured via Doppler ultrasound before and after 2 weeks of each intervention.
Forearm muscle oxygenation at rest and during rhythmic handgrip exercise with and without lower-body negative pressure | 2 weeks of each intervention
  Muscle oxygen saturation will be measured via near-infrared spectroscopy before and after 2 weeks of each intervention.

SECONDARY OUTCOMES:
Beat-to-beat blood pressure at rest and during rhythmic handgrip exercise with and without lower-body negative pressure | 2 weeks of each intervention
  Blood pressure will be measured via a finger cuff (finometer) before and after 2 weeks of each intervention.
Aortic hemodynamics at rest and during rhythmic handgrip exercise with and without lower body negative pressure | 2 weeks of each intervention
  Aortic blood pressure and pressure waves will be assessed using radial applanation tonometry before and after 2 weeks of each intervention.
Stroke volume at rest and during rhythmic handgrip exercise with and without lower body negative pressure | 2 weeks of each intervention
  Stroke volume will be assessed via impedance cardiography before and after 2 weeks of each intervention.
Heart rate at rest and during rhythmic handgrip exercise with and without lower body negative pressure | 2 weeks of each intervention
  Heart rate will be assessed via impedance cardiography before and after 2 weeks of each intervention.
Systemic vascular resistance at rest and during rhythmic handgrip exercise with and without lower body negative pressure | 2 weeks of each intervention
  Systemic vascular resistance will be assessed via impedance cardiography before and after 2 weeks of each intervention.
Central and peripheral arterial stiffness at rest | 2 weeks of each intervention
  Carotid-femoral and femoral-dorsalis pedis pulse wave velocity will be measured using arterial applanation tonometry before and after 2 weeks of each intervention.
Forearm muscle strength | 2 weeks of each intervention
  Maximal forearm muscle strength will be measured using a handgrip dynamometer before and after 2 weeks of each intervention.
L-arginine levels | 2 weeks of each intervention
  Serum levels of l-arginine will be assessed before and after 2 weeks of each intervention.
Nitric oxide levels | 2 weeks of each intervention
  Serum levels of nitric oxide will be assessed before and after 2 weeks of each intervention.
L-citrulline levels | 2 weeks of each intervention
  Serum levels of l-citrulline will be assessed before and after 2 weeks of each intervention.
L-ornithine levels | 2 weeks of each intervention
  Serum levels of l-ornithine will be assessed before and after 2 weeks of each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maharaj A, Fischer SM, Dillon KN, Kang Y, Martinez MA, Figueroa A. Acute Citrulline Blunts Aortic Systolic Pressure during Exercise and Sympathoactivation in Hypertensive Postmenopausal Women. Med Sci Sports Exerc. 2022 May 1;54(5):761-768. doi: 10.1249/MSS.0000000000002848. Epub 2022 Jan 3. PMID 34974502
- [Background] Maharaj A, Fischer SM, Dillon KN, Kang Y, Martinez MA, Figueroa A. Effects of L-Citrulline Supplementation on Endothelial Function and Blood Pressure in Hypertensive Postmenopausal Women. Nutrients. 2022 Oct 20;14(20):4396. doi: 10.3390/nu14204396. PMID 36297080
- [Background] Kang Y, Dillon KN, Martinez MA, Maharaj A, Fischer SM, Figueroa A. Combined L-Citrulline Supplementation and Slow Velocity Low-Intensity Resistance Training Improves Leg Endothelial Function, Lean Mass, and Strength in Hypertensive Postmenopausal Women. Nutrients. 2022 Dec 23;15(1):74. doi: 10.3390/nu15010074. PMID 36615732
- [Background] Figueroa A, Maharaj A, Kang Y, Dillon KN, Martinez MA, Morita M, Nogimura D, Fischer SM. Combined Citrulline and Glutathione Supplementation Improves Endothelial Function and Blood Pressure Reactivity in Postmenopausal Women. Nutrients. 2023 Mar 23;15(7):1557. doi: 10.3390/nu15071557. PMID 37049398
- [Background] Figueroa A, Alvarez-Alvarado S, Jaime SJ, Kalfon R. l-Citrulline supplementation attenuates blood pressure, wave reflection and arterial stiffness responses to metaboreflex and cold stress in overweight men. Br J Nutr. 2016 Jul;116(2):279-85. doi: 10.1017/S0007114516001811. Epub 2016 May 10. PMID 27160957